CLINICAL TRIAL: NCT05232071
Title: A Placebo-controlled, Proof-of-concept Study to Evaluate the Safety and Efficacy of Lanifibranor Alone and in Combination With the Sodium-glucose Transport Protein 2 (SGLT2) Inhibitor EmpaGliflozin in patiEnts With Non-alcoholic Steatohepatitis (NASH) and Type 2 Diabetes Mellitus (T2DM)
Brief Title: Placebo-controlled, Proof-of-concept Study to Evaluate the Safety and Efficacy of Lanifibranor Alone and in Combination With SGLT2 Inhibitor EmpaGliflozin in patiEnts With NASH and Type 2 Diabetes Mellitus
Acronym: LEGEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inventiva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 337HNAS21016
Record Dates: First submitted 2022-01-26; First posted 2022-02-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — lanifibranor; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lanifibranor (IVA337) (800 mg/day) (Experimental): 2 Lanifibranor tablets 400 mg with food --> once a day (quaque die, QD)
  Interventions: Drug: IVA337
- Matching placebo (Placebo Comparator): 2 Placebo to match tablets with food --> once a day (quaque die, QD)
  Interventions: Drug: Placebo
- Lanifibranor (IVA337) (800 mg/day) plus Empagliflozin (10mg/day) (Experimental): 2 Lanifibranor tablets 400 mg plus 1 Empagliflozin tablet 10mg with food --> once a day (quaque die, QD)
  Interventions: Drug: IVA337; Drug: Empagliflozin

INTERVENTIONS:
Drug: IVA337 — 800 mg
  Other Names: Lanifibranor
  Arms: Lanifibranor (IVA337) (800 mg/day); Lanifibranor (IVA337) (800 mg/day) plus Empagliflozin (10mg/day)
Drug: Placebo — Placebo to match
  Arms: Matching placebo
Drug: Empagliflozin — 10 mg
  Other Names: Jardiance
  Arms: Lanifibranor (IVA337) (800 mg/day) plus Empagliflozin (10mg/day)

SUMMARY:
The study in the T2DM population is intended to confirm the lanifibranor effect versus placebo on glycemic control and assess a positive effect of the combination of lanifibranor with an SGLT2 inhibitor on glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years at the time of signing informed consent
2. Diagnosis of NASH, based on histology or cT1≥875ms assessed by LiverMultiScan or cT1≥825ms assessed by LiverMultiScan and hepatic fat content ≥ 10% assessed by MRI-PDFF at screening
3. HbA1c at screening ≥ 7.0 and ≤ 10.0%, on diet alone, or on metformin and/or dipeptidyl peptidase 4 inhibitor (DPP-IVi) therapy. Both with doses to be stable for 3 months
4. Negative pregnancy test at Screening for females of childbearing potential or at least two-year post-menopausal.

Exclusion Criteria:

Liver-related:

1. Documented causes of chronic liver disease other than NASH
2. Histologically documented liver cirrhosis (fibrosis stage F4)
3. History or current diagnosis of hepatocellular carcinoma (HCC)
4. History of or planned liver transplant
5. Documented history of human immunodeficiency virus (HIV) infection
6. ALT or AST > 5 × upper limit of normal (ULN)
7. Abnormal liver function as defined by central laboratory evaluation:

   Albumin < LLN INR ≥ 1.3 (unless patient is on anticoagulants) Total bilirubin level ≥ 1.5 mg/dL (25.7 µmol/L) (patients with a documented history of Gilbert's syndrome can be enrolled if direct bilirubin is ≤ 0.45 mg/dL (7.7 μmol/L) )
8. Hemoglobin < 110 g/L (11 g/dL) for females and < 120 g/L (12 g/dL) for males
9. WBC < LLN. A lower count is acceptable in patients with benign ethnic neutropenia, if considered to be clinical insignificant by the investigator
10. Platelet count < 140,000/µL
11. ALP > 2 × ULN
12. Patient currently receiving any approved treatment for NASH or obesity
13. Current or recent history (< 5 years) of significant alcohol consumption
14. Administration of drugs known to produce hepatic steatosis in the 6 months prior to Screening.

    Diabetes related:
15. Diabetes mellitus other than type 2
16. Diabetic ketoacidosis at Screening
17. Current treatment with glucagon-like peptide-1 receptor agonists (GLP-1RA), insulin or sulfonylurea or treatment within the last 3 months prior to Screening
18. Patients on pioglitazone in the last 12 months prior to Screening.
19. Patients on metformin, DPP-IVi, thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels, unless on stable doses in last 3 months

    Obesity related:
20. BMI>45 kg/m2 at screening
21. Introduction of an anti-obesity drug or restrictive bariatric surgery in the past 12 months prior to Screening or planned bariatric surgery through Week 24.

Cardiovascular related:

21. History of or current unstable cardiac dysrhythmias 22. Unstable heart failure 23. Uncontrolled hypertension 24. Stroke or transient ischemic attack

General safety:

25. Significant systemic or major illnesses other than liver disease and pulmonary disease, organ transplantation, serious psychiatric disease, that, in the opinion of the investigator, would preclude treatment with lanifibranor and/or adequate follow up 26. Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value < 60 mL/min 27. Concomitant treatment with PPAR-⍺ agonists (fibrates) 28. Patients on Vitamin E at doses ≥ 400 IU/day; doses of ≥ 400 IU/day are allowed when no qualitative change in dose for 6 months prior to Screening 29. Have a known hypersensitivity to any of the IMPs 30. Previous exposure to lanifibranor or empagliflozin 31. Present pregnancy/lactation 32. Metallic implant of any sort that prevents MRI examination 33. Participation in any clinical trial of an approved or non approved investigational medicinal product/device within 3 months from Screening or five half-lives of the investigational drug from Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Assessment of the effect of lanifibranor alone compared to placebo and the effect of lanifibranor in combination with empagliflozin compared to placebo on absolute change in HbA1c from baseline (Week 0) to Week 24 | Date of randomisation until the end of treatment at week 24
  Absolute change in HbA1c from baseline (Week 0) to Week 24

CONTACTS AND LOCATIONS:
Locations (42):
- United States (26):
  - Birmingham Digestive Health Research, Homewood, Alabama
  - Institute for Liver Health dba Arizona Liver Health, Chandler, Arizona
  - ARcare Center for Clinical Research, Conway, Arkansas
  - ARcare Center for Clinical Research, Little Rock, Arkansas
  - Cure Clinical Research, LLC, Fountain Valley, California
  - Velocity Clinical Research, Gardena, California
  - National Research Institute, Huntington Park, California
  - Cadena Care Institute, LLC, Poway, California
  - Florida Research Institute, Lakewood Rch, Florida
  - Galenus Group, Lehigh Acres, Florida
  - Prolive Medical Research, Miami, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Digestive Health Research of Southern California, South Bend, Indiana
  - Tandem Clinical Research - New Orleans Area Site, Marrero, Louisiana
  - Harvard Medical School, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - AIG Digestive Disease Research, Florham Park, New Jersey
  - Digestive Health Research, Hermitage, Tennessee
  - Accelemed Research Institute, Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - American Research Corporation, San Antonio, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Impact Research Institute, Waco, Texas
  - Digestive Health Research of North Texas, Wichita Falls, Texas
  - University of Virginia, Charlottesville, Virginia
  - Central Virginia VA Healthcare System, Richmond, Virginia
- Belgium (5):
  - CUB Erasme Hospital, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - UZ GENT, Ghent
- France (6):
  - CHU Angers_Service d'hepatogastro-enterologie, Angers
  - CHU Limoges, Limoges
  - Hopital Saint Antoine, Paris
  - CHU Bordeaux, Pessac
  - Chu Rangueil, Toulouse
  - HGE CHRU Nancy, Vandœuvre-lès-Nancy
- Amsterdam UMC, Amsterdam, Netherlands
- United Kingdom (4):
  - Hull University Teaching Hospital, Hull
  - King's College Hospital, London
  - St Georges Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne